CLINICAL TRIAL: NCT06007040
Title: Interstitial Lung Disease Associated
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-PCCM-ILD
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Interstitial Lung Disease
Keywords: Interstitial lung disease, ANCA, CTD, IPAF, IIP
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This single-center, retrospective cohort study was conducted to determine whether ANCA-ILD spectrum share the same clinical manifestations and outcome with CTD feature disease spectrum.

DETAILED DESCRIPTION:
We retrospectively reviewed patients who had been diagnosed with interstitial pneumonia during outpatient or hospitalization at Peking Union Medical College Hospital (PUMCH) between January 2012 and December 2021.

1. Baseline data collection:

   1. Baseline information at the time of initial diagnosis was obtained, and the following items were analyzed: demographic information (age, gender), clinical course, clinical symptoms and signs, laboratory findings [routine blood, erythrocyte sedimentation rate (ESR), hypersensitivity C-reactive protein (Hs-CRP), rheumatoid factor (RF) and serologic autoantibodies], pulmonary function tests (PFTs), and chest HRCT scans.
   2. MPO-ANCA and PR3-ANCA titers were measured by ELISA.
   3. Chest HRCT images were evaluated by at least two pulmonologists and radiologists. The HRCT scans were analyzed for the following characteristics: ground-glass opacities, reticular patterns, honeycombing, traction bronchiectasis.
   4. Spirometry was performed according to standardized guidelines. PFTs results were expressed as percentages of the predicted values, thereby correcting for age, gender and bodyweight.
2. Treatment was defined as the use of corticosteroids ≥ 10mg/d, azathioprine, cyclophosphamide, mycophenolate mofetil, methotrexate, or rituximab. Follow-up was up to the time of patient's last visit or time of death, and the outcomes were defined as death from all causes.
3. Outcome

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Aged from 18 to 85 years with informed consent
* Have a diagnosis of ILD based on clinical symptoms and radiologic features, with or without histopathologic results

Exclusion Criteria:

* ILD induced by drug, environment, or occupational exposure
* Hypersensitivity pneumonitis and sarcoidosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Interstitial pneumonia based on clinical symptoms and radiologic features, with or without histopathologic results.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | From baseline until the date of death from all cause, up to 5 years
  death from all causes

CONTACTS AND LOCATIONS:
Overall Officials: Juhong Shi, M.D, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No